CLINICAL TRIAL: NCT02395198
Title: Epidemiology of Hepatitis C Virus Infection Among Opioid Substituted Patients: Factors Influencing Treatment Initiation and Seroconversion
Brief Title: Epidemiology of Hepatitis C Virus Infection Among Opioid Substituted Patients
Acronym: ECHO
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Prof. Dr. med. Jens Reimer (Other)
Collaborators: Janssen-Cilag G.m.b.H (Industry)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. Jens Reimer, Head, Addiction Medicine Unit, University Medical Center Hamburg Eppendorf; Centre for Interdisciplinary Addiction Research (CIAR), Hamburg University, Universitätsklinikum Hamburg-Eppendorf
Organization: Universitätsklinikum Hamburg-Eppendorf (Other)
Other Study IDs: 12748
Record Dates: First submitted 2015-03-16; First posted 2015-03-23 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Hepatitis C
Keywords: hepatitis c virus; opioid substitution treatment
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HCV negative or in HCV treatment at T1: This group will be followed up at T2

SUMMARY:
The aim of the present study is to estimate the national annual prevalence and incidence of current hepatitis C virus (HCV) infections among opioid dependent individuals in opioid substitution treatment (OST) based on a representative sample of approximately 2,500 outpatients in 100 substitution facilities across Germany. Furthermore, the study aims to describe factors influencing HCV therapy initiation and seroconversion during OST.

DETAILED DESCRIPTION:
In this non-interventional, observational, longitudinal study, data is collected at two time points. The primary outcome measures HCV prevalence and incidence will be based on documentation from routine patient care at baseline and 12-month follow-up. Secondary outcome measures will be investigated by means of surveys of opioid substituted patients and their clinicians (completed at baseline), as well as data from routine patient care.

The sample size calculation is based on the primary outcome variable of HCV incidence among OST patients. The literature reports an HCV incidence of about 4/100 person-years +/- 2 new infections per 100 person-years in this target group. For a partial sample size of (at least) 32 patients with HCV seroconversion and an observation period of 1 year, 800 HCV antibody-negative patients are needed as an initial group for observation. Assuming an HCV antibody prevalence of 68% among OST patients, 2500 patients are needed in total (32% corresponds to N = 800).

Recruitment of clinicians is conducted via the national Substitution Registry in which all clinicians in Germany, who hold a qualification to prescribe substitution medication, are registered. To ensure that all substituting clinicians in Germany are considered in the present study, the investigators sent study invitations to all 3,356 addresses in the Substitution Registry as of 31.12.2013. Of the clinicians eligible for participation, a representative sample of clinician is drawn according to two criteria: 'German Federal State' (GFS) and 'Number of Patients Per Clinician' (PPC). Using the SPSS Complex Samples Procedure, clinicians are stratified by GFS and PPC, such that each GFS is represented at least once, and such that the same proportions of clinicians per GFS and per PPC category are achieved (to the best of our ability) as in the total sample of clinicians registered in the Substitution Registry.

ELIGIBILITY:
Inclusion Criteria:

* minimum age 18
* diagnosed opioid dependence according to the ICD-10
* currently in opioid substitution treatment

Exclusion Criteria:

* severe mental impairment
* insufficient German reading and writing skills

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Opioid dependent outpatients in opioid substitution treatment regardless of treatment setting
Sampling Method: Probability Sample
Enrollment: 2467 (Actual)
Dates: Start 2014-08; Primary Completion 2017-04 (Actual); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
National annual prevalence and incidence of current HCV infections among opioid dependent individuals in substitution treatment | 12 months

SECONDARY OUTCOMES:
Patient questionnaire: Patient Reported Outcomes | 1 month
  Quality of Life, Health-Related Quality of Life (SF-12), Physical health (OTI), Mental health (BSI-18), Autonomy preference (API-Dm), Satisfaction with care (ZAPA), Knowledge, needs and attitudes towards infectious diseases, HCV treatment and treatment experiences
Clinician questionnaire: Clinician Reported Outcomes and Data from Routine Patient Care | 1 month
  Substitution treatment, HCV diagnostic and treatment, Consumption of substances, Physical and mental health (Checklist of somatic and psychiatric diseases, CGI), Patient wellbeing (Problem severity, GAF)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Reimer, Prof. Dr., Principal Investigator — University Medical Center Hamburg-Eppendorf, Centre for Interdisciplinary Addiction Research (CIAR), Hamburg University
Locations (32):
- Germany (32):
  - Dr. Rudolf Dinkelacker, Crailsheim, Baden-Wurttemberg
  - Dr. Manfred Hartmann, Herrenberg, Baden-Württenberg
  - Dr. Reinhold Burr, Hirrlingen, Baden-Württenberg
  - Dr. Christoph von Ascheraden, Saint Blasien, Baden-Württenberg
  - Dr. Barbara Haider, Aichach, Bavaria
  - Dr. Eugen Fürmann, Augsburg, Bavaria
  - Dr. Astrid Beck, Fürstenfeldbruck, Bavaria
  - Dr. Winfred Dresel, Warngau, Bavaria
  - Dr. Monika Peter-Giglio, Bad Nauheim, Hesse
  - Dr. Andreas Weselek, Ehringshausen, Hesse
  - Dr. Georg Wetzig, Frankfurt am Main, Hesse
  - Dr. Christine Rose, Goslar, Lower Saxony
  - Dr. Uta Menschikowski, Parchim, Mecklenburg-Vorpommern
  - Dr. Georg Kramann, Achim, Niedersachen
  - Dr. Detmar Jobst, Bonn, North Rhine-Westphalia
  - Dr. Michel Voss, Cologne, North Rhine-Westphalia
  - Dr. Helmut Walter, Hamm, North Rhine-Westphalia
  - Dr. Manfred Plum, Herne, North Rhine-Westphalia
  - Dr. Martin Burger und Dr. Wolfgang Lüttecken, Münster, North Rhine-Westphalia
  - Dr. Astrid Weber, Koblenz, Rhineland-Palatinate
  - Dr. Liane Arimond, Trier, Rhineland-Palatinate
  - Dr. Maria Viehweger, Chemnitz, Saxony
  - Dr. Ernst Soldan, Norderstedt, Schleswig-Holstein
  - Dr. Alexander Cegla, Wenningstedt, Schleswig-Holstein
  - Dr. Gerd Klausen, Berlin
  - Dr. Clemens Micus, Berlin
  - Dr. Lutz Weinrich, Berlin
  - Dr. Wieland Tietje, Bremen
  - Dr. Nico le Claire, Hamburg
  - Dr. Felix Maas, Hamburg
  - Dr. Wirkner Thiel, Hamburg
  - Dr. Eckhard Zeigert, Hamburg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Strada L, Schmidt CS, Rosenkranz M, Verthein U, Scherbaum N, Reimer J, Schulte B. Factors associated with health-related quality of life in a large national sample of patients receiving opioid substitution treatment in Germany: A cross-sectional study. Subst Abuse Treat Prev Policy. 2019 Jan 3;14(1):2. doi: 10.1186/s13011-018-0187-9. PMID 30606188
- [Derived] Strada L, Schulte B, Schmidt CS, Verthein U, Cremer-Schaeffer P, Kruckeberg S, Reimer J. Epidemiology of hepatitis C virus infection among people receiving opioid substitution therapy (ECHO): study protocol. BMC Infect Dis. 2015 Dec 10;15:563. doi: 10.1186/s12879-015-1307-z. PMID 26653754